CLINICAL TRIAL: NCT04593602
Title: Early Mobilization in Older Adults With Acute Cardiovascular Disease: A Prospective, Multi-centre Stepped Wedge Cluster Randomized Trial
Brief Title: Early Mobilization in Older Adults With Acute Cardiovascular Disease
Acronym: EM-HEART
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Changed research approach
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Clinician-Investigator, Lady Davis Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Lady Davis Institute
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Early Mobilization; Older Adults; Acute Cardiovascular Disease; Nursing
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: In the stepped-wedge cluster design, there is random and sequential crossover of clusters from control (phase 1) to intervention (phase 2) until all clusters are exposed. The nature of the intervention requires randomization of entire units to the intervention with associated mobility culture change and this precludes a standard randomized controlled trial design (i.e., randomization of some patients to the intervention but not others). The stepped-wedge design allows each site to function as its own control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Mobilization Intervention (Experimental): The bedside nurse determines the prehospital Level of Function based on patient and family report and current Level of Function based on nursing mobility assessment. Each Level of Function has 3 primary activities designed to promote the patient to the next level. The nurse leads mobility activities based on the patient's current Level of Function once per shift, twice daily (AM+PM). If a patient is able to complete each of the 3 activities, the nurse on the subsequent shift will assess whether the Level of Function can be advanced. Physiotherapy consultation is available if required, although not obligatory. Patients are encouraged to spend as much time in the chair and ambulatory as possible.
  Interventions: Behavioral: Early Mobilization
- Usual Mobility Care (Active Comparator): Usual mobility care involves following physician orders for mobilization (i.e., bedrest, mobilization to chair with meals, physiotherapy consultation and care) as per local practice.
  Interventions: Behavioral: Usual Mobility Care

INTERVENTIONS:
Behavioral: Early Mobilization — Nurse-driven early mobilization activities twice daily
  Arms: Early Mobilization Intervention
Behavioral: Usual Mobility Care — Usual mobility care involves following physician orders for mobilization (i.e., bedrest, mobilization to chair with meals, physiotherapy consultation and care) as per local practice.
  Arms: Usual Mobility Care

SUMMARY:
The EM-HEART study is a prospective, multi-centre stepped wedge cluster randomized trial to evaluate the effectiveness of a pragmatic early mobilization (EM) program to improve patient-centred and clinical outcomes in older adults with acute CV disease. There will be 256 participants ≥60 years old with acute CV disease enrolled at 6 participating Canadian hospitals. The study will investigate whether EM improves functional status during admission, as compared to usual care, and whether this leads to improved health-related quality of life post-hospitalization. Functional status will be measured with the validated Level of Function Mobility Scale. The primary outcome will be the Short-Form SF-36 physical component scale score at 1-month post-hospitalization. Secondary outcomes include functional status and hospital readmission at 1-month post-hospitalization.

DETAILED DESCRIPTION:
The EM-HEART study is a prospective, multi-centre stepped wedge cluster randomized trial to evaluate the effectiveness of a pragmatic EM program to improve patient-centred and clinical outcomes in older adults with acute CV disease. There will be 256 participants ≥60 years old with acute CV disease enrolled at 6 participating Canadian hospitals. The study will investigate whether EM improves functional status during admission, as compared to usual care, and whether this leads to improved health-related quality of life post-hospitalization. Functional status will be measured with the validated Level of Function Mobility Scale. The primary outcome will be the Short-Form SF-36 physical component scale score at 1-month post-hospitalization. Secondary outcomes include functional status and hospital readmission at 1-month post-hospitalization. Nested cohort studies will explore (1) the relationship between EM, sedentary time, and posthospitalization outcomes and (2) the impact of EM on muscle mass loss and inflammation in older adults with acute CV disease.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* no planned cardiac surgery during admission

Exclusion Criteria:

* projected cardiac ICU stays less than 24 hours
* patients unable to complete follow-up

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Short Form (SF)-36 Physical Component Summary (PCS) score at 1-month post-hospitalization | 1 month post-hospitalization
  Health-related quality of life

SECONDARY OUTCOMES:
SF-36 Physical Component Scale score | 12 months post-hospitalization
  Health-related quality of life
SF-36 Mental Component Summary score | 1 month post-hospitalization
  Health-related quality of life
SF-36 Mental Component Summary score | 12 months post-hospitalization
  Health-related quality of life
Level of Function Mobility Score | 1 month post-hospitalization
  Functional status
Level of Function Mobility Score | 12 months post-hospitalization
  Functional status
Hospital readmission | 1 month post-hospitalization
  Resource use outcome
Hospital readmission | 12 months post-hospitalization
  Resource use outcome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Semsar-Kazerooni K, Dima D, Valiquette J, Berube-Dufour J, Goldfarb M. Early Mobilization in People With Acute Cardiovascular Disease. Can J Cardiol. 2021 Feb;37(2):232-240. doi: 10.1016/j.cjca.2020.03.038. Epub 2020 Apr 2. PMID 32739452